CLINICAL TRIAL: NCT03701074
Title: Single Center, Randomized, Double Blind, Placebo Controlled Trial to Evaluate the Safety and Efficacy of Acetaminophen in Preterm Infants Used in Combination With Ibuprofen for Closure of the Ductus Arteriosus
Brief Title: Randomized Controlled Trial to Evaluate the Safety and Efficacy of Acetaminophen in Preterm Infants Used in Combination With Ibuprofen for Closure of the Ductus Arteriosus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: very slow enrollment. Only one patient enrolled. Termination by PI
Sponsor: University of South Alabama (Other)
Responsible Party: Principal Investigator, Ramachandra Bhat, Assistant Professor, University of South Alabama
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-081/730216-8
Record Dates: First submitted 2018-08-22; First posted 2018-10-09 (Actual); Results first posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: Patent Ductus Arteriosus; Preterm Infant; Bronchopulmonary Dysplasia
Keywords: patent ductus arteriosus; acetaminophen; ibuprofen; bronchopulmonary dysplasia; mechanical ventilation
MeSH Terms: conditions — Ductus Arteriosus, Patent; Premature Birth; Bronchopulmonary Dysplasia | interventions — Ibuprofen; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ibuprofen and acetaminophen arm (intervention arm) (Experimental): ibuprofen and acetaminophen will be administered concomitantly. Ibuprofen will be administered through intravenous route. The dose of ibuprofen will be the standard dosing regimen used in our unit: dosing based on the postnatal age. For Infants > 108 h of postnatal age: 18 mg/kg/dose loading dose followed by 9 mg/kg/dose, two doses at q24 intervals, started 24 h after the loading dose. Acetaminophen will be administered as oral formulation. Acetaminophen is given at a dose of 15 mg/Kg/dose, q 6 hours, for 3 days (total of 12 doses).
  Interventions: Drug: Ibuprofen and acetaminophen
- ibuprofen and placebo arm (control arm) (Active Comparator): ibuprofen and acetaminophen will be administered concomitantly. Ibuprofen will be administered through intravenous route. The dose of ibuprofen will be the standard dosing regimen used in our unit: dosing based on the postnatal age. For Infants > 108 h of postnatal age: 18 mg/kg/dose loading dose followed by 9 mg/kg/dose, two doses at q24 intervals, started 24 h after the loading dose. Placebo will be sterile water, with similar volume and color as acetaminophen, will be given through the oro-gastric tube, for three days at 6 h intervals.
  Interventions: Drug: Ibuprofen and placebo

INTERVENTIONS:
Drug: Ibuprofen and acetaminophen — Intravenous ibuprofen given concomitantly with oral acetaminophen
  Arms: ibuprofen and acetaminophen arm (intervention arm)
Drug: Ibuprofen and placebo — Intravenous ibuprofen given concomitantly with oral placebo
  Arms: ibuprofen and placebo arm (control arm)

SUMMARY:
The purpose of the present study is to determine whether treatment of hemodynamically significant patent ductus arteriosus with a combined therapy of intravenous Ibuprofen and oral acetaminophen has higher success rate in closing the ductus arteriosus than a standard treatment strategy of using intravenous ibuprofen alone among preterm infants.

DETAILED DESCRIPTION:
The primary objectives of the study are to confirm the safety of oral acetaminophen in extremely low birth infants, given concomitantly with intravenous ibuprofen and also to determine its efficacy in significantly increasing the rates of ductal closure when compared to only intravenous ibuprofen therapy. Hence primary outcome variable include patent ductus arteriosus closure success rate, based on the 2-D transthoracic echocardiographic evidence.

This study is a single center, randomized, double blinded, placebo controlled trial. Preterm infants with gestational age of with a gestational age ≤27 6/7 weeks by the best obstetric estimate are eligible for enrollment.

For randomization, the study population will be stratified to two subgroups based on gestational age (GA ≤24 weeks and > 25 weeks). Randomization will occur by using computer generated random sequence, using a 4-block design, with 1:1 parallel allocation. Allocations include treatment and control arm. Treatment arm will receive combination of intravenous ibuprofen and oral acetaminophen, while control arm will receive intravenous Ibuprofen and oral placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Preterm infant ≤27 6/7
2. Written parental consent is obtained
3. Infant requires respiratory support
4. diagnosis of a persistent patent ductus arteriosus after 5 days of age, (defined as at least two of the following:

   1. Ductus size ≥ 1.5 mm
   2. Maximum flow velocity through the ductus ≤ 2 m/s
   3. Left atrium to aorta ratio ≥ 1.4
   4. Wide pulse pressure
   5. B-type natriuretic peptide (BNP)
5. Attending neonatologist made decision to treat patent ductus arteriosus

Exclusion Criteria:

1. No parental consent
2. Infants > 21days of postnatal age
3. Congenital anomalies such as cardiac or multiple anomalies
4. Infection (e.g., septicemia, pneumonia)
5. Bleeding disorder or platelet count< 50,000/ml
6. Acute kidney injury (AKI)defined as oliguria (urine output< 0.5 ml/kg/hr for 16hrs) and/or serum creatinine > 1.5 mg/dl
7. Elevated liver enzymes (>2 fold from upper normal limits)
8. Pulmonary hypertension or right to left shunt through the ductus arteriosus
9. Diagnosis of necrotizing enterocolitis
10. Unable to tolerate oral medications at the time of enrollment.

Ages: 5 Days to 21 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fabien Eyal, MD, Study Director — University of South Alabama
Locations (1):
- University of South Alabama, Mobile, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall screening for the study enrollment started 12/15/2018. Screening was continued until 10/30/2020. The study was conducted at the Neonatal Intensive Care Unit
Groups:
- Ibuprofen and Placebo Arm (Control Arm): ibuprofen and placebo will be administered concomitantly. Ibuprofen will be administered through intravenous route. The dose of ibuprofen will be the standard dosing regimen used in our unit: dosing based on the postnatal age. For Infants > 108 h of postnatal age: 18 mg/kg/dose loading dose followed by 9 mg/kg/dose, two doses at q24 intervals, started 24 h after the loading dose. Placebo will be sterile water, with similar volume and color as acetaminophen, will be given through the oro-gastric tube, for three days at 6 h intervals.
  Ibuprofen and placebo: Intravenous ibuprofen given concomitantly with oral placebo
Period: Overall Study
Arm/Group | Ibuprofen and Acetaminophen Arm (Intervention Arm) | Ibuprofen and Placebo Arm (Control Arm)
Started | 1 | 0
Completed | 0 (Treatment was withdrawn after the 10th dose of oral medication (acetaminophen), on day 3 of treatment, as the infant developed mild abdominal distension which was as per the study protocol) | 0
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Overall only one infant was enrolled into the study. Hence, control arm had no patient enrolled
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibuprofen and Acetaminophen Arm (Intervention Arm) | Ibuprofen and Placebo Arm (Control Arm) | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 1 |  | 1
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1
PDA size [Number; unit: mm] | 1.5 |  | 1.5

OUTCOME MEASURES:

1. Primary Outcome: Ductus Arteriosus Closure/Constriction Rate
Description: Ductal closure/constriction rate as defined based on the echocardiographic findings. Ductal closure/constriction will be defined as the complete closure of ductus or ductal diameter <1 mm
Time Frame: 24-48 hours after the completion of study intervention
Population: None were enrolled for the control arm
Measure: Count of Participants; unit: Participants
Arm/Group | Ibuprofen and Acetaminophen Arm (Intervention Arm) | Ibuprofen and Placebo Arm (Control Arm)
Number analyzed (Participants) | 1 | 0
Participants | 0 | 0

2. Secondary Outcome: Echocardiographic Patent Ductus Arteriosus Parameters Before and After the Study Intervention
Time Frame: 24-48 hours after the completion of study intervention
Reporting Status: Not Posted

3. Secondary Outcome: Ventilatory Settings Before and After the Study Intervention
Time Frame: 24-48 hours after the completion of study intervention
Reporting Status: Not Posted

4. Secondary Outcome: Rate of Liver Injury
Description: liver enzymes before and after the study intervention
Time Frame: 24-48 hours after the completion of study intervention
Reporting Status: Not Posted

5. Secondary Outcome: Rate of Renal Injury
Description: Blood urea nitrogen (BUN) and serum creatinine before and after the study intervention
Time Frame: 24-48 hours after the completion of study intervention
Reporting Status: Not Posted

6. Secondary Outcome: Rate of Hematological Adverse Events
Description: Hematocrit and platelets before and after the study intervention
Time Frame: 24-48 hours after the completion of study intervention
Reporting Status: Not Posted

7. Secondary Outcome: Total Number of Days of Mechanical Ventilation
Time Frame: from randomization until discharge/40 weeks post menstrual age
Reporting Status: Not Posted

8. Secondary Outcome: Total Number of Days of Need for Supplemental Oxygen
Time Frame: from randomization until discharge/40 weeks post menstrual age
Reporting Status: Not Posted

9. Secondary Outcome: Duration of Noninvasive Ventilation
Time Frame: from randomization until discharge/40 weeks post menstrual age
Reporting Status: Not Posted

10. Secondary Outcome: Rate of Persistence of Ductus-needing Pharmacological Treatment
Time Frame: from randomization until discharge/40 weeks post menstrual age
Reporting Status: Not Posted

11. Secondary Outcome: Rate of Surgical Ligation of PDA
Time Frame: from randomization until discharge/40 weeks post menstrual age
Reporting Status: Not Posted

12. Secondary Outcome: Rate of Bronchopulmonary Dysplasia
Time Frame: at 36 weeks post menstrual age
Reporting Status: Not Posted

13. Secondary Outcome: Percentage of Infants Requiring Home Oxygen Therapy
Time Frame: at discharge/40 weeks post menstrual age
Reporting Status: Not Posted

14. Secondary Outcome: Death Before Discharge
Time Frame: until discharge/40 weeks post menstrual age
Reporting Status: Not Posted

15. Secondary Outcome: Time to Achieve Full Enteral Feeding
Description: Time to achieve 120 ml/kg/day of enteral feeding
Time Frame: from birth until discharge/40 weeks post menstrual age
Reporting Status: Not Posted

16. Secondary Outcome: Days on Total Parenteral Nutrition
Time Frame: from birth until discharge/40 weeks post menstrual age
Reporting Status: Not Posted

17. Secondary Outcome: Retinopathy of Prematurity
Time Frame: from birth until discharge/40 weeks post menstrual age
Reporting Status: Not Posted

18. Secondary Outcome: Rate of Spontaneous Intestinal Perforation
Time Frame: from randomization until discharge/40 weeks post menstrual age
Reporting Status: Not Posted

19. Secondary Outcome: Rate of Necrotizing Enterocolitis
Time Frame: from randomization until discharge/40 weeks post menstrual age
Reporting Status: Not Posted

20. Secondary Outcome: Rate of Gastrointestinal Hemorrhage
Time Frame: from randomization until discharge/40 weeks post menstrual age
Reporting Status: Not Posted

21. Secondary Outcome: Rate of Late Onset Sepsis
Time Frame: from randomization until discharge/40 weeks post menstrual age
Reporting Status: Not Posted

22. Secondary Outcome: Length of Hospital Stay
Time Frame: from birth until discharge/40 weeks post menstrual age
Reporting Status: Not Posted

23. Secondary Outcome: Rate of Periventricular Leukomalacia
Time Frame: from randomization until discharge/40 weeks post menstrual age
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 4 months
Description: None were enrolled into control arm, Therefore, number infants at risk for adverse events under the control arm are zero
Arm/Group | Ibuprofen and Acetaminophen Arm (Intervention Arm) | Ibuprofen and Placebo Arm (Control Arm)
All-Cause Mortality (participants affected / at risk) | 1/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ibuprofen and Acetaminophen Arm (Intervention Arm) (N=1) | Ibuprofen and Placebo Arm (Control Arm) (N=0)
Biochemical evidence of acute kidney injury with preserved renal function, probably nor related to i (Renal and urinary disorders) | 1 | 0 — As per the study protocol, after the completion of study intervention, kidney function was monitored using BUN and serum creatinine. S. creatinine was noted to be 2 times above the baseline pre-intervention level (1.28 mg/dl). Renal function normal

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-07): https://cdn.clinicaltrials.gov/large-docs/74/NCT03701074/Prot_SAP_000.pdf